CLINICAL TRIAL: NCT03620487
Title: Pathogen Detection and Host Response in Plasma of Patients With Dengue and Dengue Fever Like Illnesses in Nepal.
Brief Title: Detection of Dengue Virus in Plasma of Patients in Nepal
Status: Completed | Type: Observational
Sponsor: Karius, Inc. (Industry)
Collaborators: Tribhuvan University, Nepal (Other)
Responsible Party: Sponsor
Other Study IDs: 012-DL-01
Record Dates: First submitted 2018-05-11; First posted 2018-08-08 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Dengue Fever
Keywords: NGS; Sequencing
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma

SUMMARY:
To test whether Karius Infectious Disease Diagnostic Sequencing assay can detect Dengue Virus in plasma from suspected cases of Dengue or Dengue Fever like-illnesses from samples collected as part of a hospital-based multi-site study conducted in Nepal.

DETAILED DESCRIPTION:
Blood samples will be obtained from consented subjects as part of a hospital-based multi-site study conducted in Nepal and will be shipped to Karius, Redwood City, CA.

The investigators will test whether the Karius test can detect Dengue Virus in plasma from those suspected cases and measure the performance of the Karius test against standard tests (PCR, ELISA test and neutralization assays) used to determine a final diagnosis of Dengue Fever.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older, suspected of having Dengue or Dengue Fever-like illnesses.

Exclusion Criteria:

* Inability to understand instructions and comply with study-related procedures, inability to understand and/or sign informed consent, any condition that will prevent the subject from completing the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with Dengue or Dengue Fever-like illnesses in Nepal.
Sampling Method: Non-Probability Sample
Enrollment: 643 (Actual)
Dates: Start 2016-10-26 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity of the Karius Test in detecting the Dengue Virus in plasma. | 3 years
  Test the sensitivity and specificity of the Karius Infectious Disease Diagnostic Sequencing Assay in detecting the Dengue Virus in plasma (measured in molecules per mL) from suspected cases of Dengue Virus from a hospital-based multicentered study conducted in Nepal.

CONTACTS AND LOCATIONS:
Overall Officials: Krishna Manandhar, PhD, Principal Investigator — Tribhuvan University
Locations (1):
- Tribhuvan University, Ki̇̄rtipur, Nepal